CLINICAL TRIAL: NCT01542164
Title: Calcium Intake and Fat Excretion - an Observational Study
Brief Title: Calcium Intake and Fat Excretion
Acronym: KIFU/B266
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Arla Foods (Industry); The Danish Dairy Research Foundation, Denmark (Other)
Responsible Party: Principal Investigator, Arne Astrup, Department of Human Nutrition, University of Copenhagen
Other Study IDs: H-B-2009-071
Record Dates: First submitted 2010-05-26; First posted 2012-03-02 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Fat Excretion; Energy Excretion
Keywords: Calcium intake; Fat excretion; Energy excretion; Gut micro flora

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, urine and faeces
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall purpose of this study is to examine the effect of calcium on fecal fat and energy excretion.

DETAILED DESCRIPTION:
Several reports have found inverse associations between calcium intake and body weight. Few intervention studies have shown that a high calcium diet resulted in a greater body weight loss than a low calcium diet. The mechanism is not clear, but one possible explanation is reduced absorption of fat in the gut, due to formation of insoluble calcium fatty acid soaps or binding of bile acids which impairs the formation of micelles.

The aim of this study is to examined for an association between habitual calcium intake and fecal energy and fat excretion, concentrations of substrates involved in energy metabolism, blood pressure and body weight

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 50 years
* healthy
* weight stable within 4 months prior to the inclusion

Exclusion Criteria:

* pregnant or lactating
* uses cholesterol lowering drugs
* on diet
* suffering from, now or previously, any gastrointestinal diseases
* elite athletes
* participation in other concomitant trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Copenhagen and Sjælland
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Total fat and energy excretion | 5 days
  Total fat and energy excretion in faeces during the test period of 5 consecutive days

SECONDARY OUTCOMES:
p-vitamin D | 1 day
p-PTH | 1 day
  Parathyroid hormone (PTH)
Selected genetic variations | 1 day
  DNA from blood sample
Blood lipids and cholesterol | 1 day
  Total p-cholesterol, p-LDL, p-HDL, p-TG and p-FFA
calcium excretion | 2 days
  Total calcium excretion in faeces and urin during the test period of 2 consecutive days
Gut micro flora | 1 day
  Identification of gut micro flora
NMR-spectroscopy based metabonomics profiling of urin | 1 day
  NMR-spectroscopy based metabonomics profiling of each test subject
blood pressure | 1 day
  Resting blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Lesli H. Larsen, Ass. Prof., Principal Investigator — Dept. of Human Nutrition, Faculty of Life Sciences, Univerity of Copenhagen
Locations (1):
- Dept. of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Frederiksberg, Copenhagen, Denmark